CLINICAL TRIAL: NCT06838897
Title: Association Between Preoperative Pain Catastrophizing Scale and Intraoperative Analgesia Consumption in Elective Laparoscopic Cholecystectomy
Brief Title: Preoperative Pain Catastrophizing and Intraoperative Analgesia Consumption
Status: Completed | Type: Observational
Sponsor: Ahmet Pece (Other)
Responsible Party: Sponsor-Investigator, Ahmet Pece, Research fellow, Samsun University
Organization: Samsun University (Other)
Other Study IDs: ceyla kolesistektomi
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Catastrophizing Pain; Pain
Keywords: pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing laparoscopic cholecystectomy

SUMMARY:
This observational study aims to evaluate the relationship between the Pain Catastrophizing Scale (PCS) and intraoperative analgesia consumption in patients undergoing laparoscopic cholecystectomy. During the preoperative period, patients will complete the Pain Catastrophizing Scale, the Beck Depression Inventory, and the Beck Anxiety Scale. During the intraoperative period, analgesia nociceptive index (ANI) electrodes will be placed, and remifentanil dosing will be adjusted accordingly. The correlation between preoperative Pain Catastrophizing Scale scores and intraoperative remifentanil consumption will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA scores of I-III
* Patients with Turkish literacy skills.
* Patients scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patients unwillingness to participate in the study.
* Conversion of surgery from laparoscopic to open surgery.
* Patients undergoing emergency laparoscopic cholecystectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective laparoscopic cholecystectomy.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanyl requirement | Intraoperative period
  The main purpose of this study is to evaluate the correlation between preoperative Pain Catastrophizing Scale and intraoperative analgesia consumption.Intraoperative analgesic dose is adjusted according to the analgesia nociceptive index.

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | up to 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale in which a respondent selectsand its correlation with the preoperative PCS score will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Üniversitesi Eğitim Ve Araştırma Hastanesi, Samsun, ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No